CLINICAL TRIAL: NCT03184103
Title: Clinical Spectrum and Outcome of Acute Post Streptococcal Glomerulonephritis in Children .
Brief Title: Acute Post Streptococcal Glomerulonephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MSHEid, Principal Investigator, Assiut University
Other Study IDs: APSGN
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: PSGN - Post-Streptococcal Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: anti streptolysin o titre and serum complement test — diagnostic lab test

SUMMARY:
Acute post streptococcal glomerulonephritis is an immunologic response of the kidney to infection, characterized by the sudden appearance of edema, hematuria, proteinuria and hypertension . It is essentially a disease of childhood that accounts for approximately 90% of renal disorders in children. The disease occurs especially in children between the ages of 2 and 12 years and young adults, and more often in male than in female .

DETAILED DESCRIPTION:
Acute post streptococcal glomerulonephritis are caused by group A beta haemolytic streptococci and follow upper airway infections such as pharyngitis or tonsillitis, by 14 to 21 days and 3-6 weeks after skin infection especially in warmer climates .

In recent decades the number of patients with post streptococcal glomerulonephritis has decreased considerably in the United States and Europe industrialized countries. In other parts of the world ,some developing communities. the incidence of post streptococcal glomerulonephritis has remained high. post streptococcal glomerulonephritis is one of the leading cause requiring hospital admissions in children , and it is also an important cause of acute renal failure in developing countries. Though deaths due to this disease are rare, it can cause serious complications such as hypertensive emergency, congestive cardiac failure, renal failure, encephalopathy and retinopathy .

Acute post streptococcal glomerulonephritis can also progress to rapidly progressive glomerulonephritis which is defined as''a syndrome that progresses rapidly within a few weeks or months to renal failure and is accompanied by urinary findings of nephritis.'' The clinical concept of rapidly progressive glomerulonephritis includes various renal diseases that cause renal function to deteriorate over a subacute course. Necrotizing crescentic glomerulonephritis is often observed in histopathological findings .

Acute post streptococcal glomerulonephritis was diagnosed in the presence of :

features of acute nephritic syndrome. evidence of recent streptococcal infection. lower serum complement three levels. Anti streptolysin o titre >200 units/ml was considered as evidence of recent streptococcal infection

ELIGIBILITY:
Inclusion Criteria:

* Children in the age groups of 2-15 years. presenting with clinical manifestation of acute nephritic syndrome will be included in the study.

Exclusion Criteria:

* Children having history suggestive of chronic renal and cardiac disease in the past
* Children with congenital renal anomalies .
* Children with clinical manifestation of nephrotic syndrome .
* Children with clinical manifestation of acute nephritic syndrome due to other causes .

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be done on children attending at Assiut University Children Hospital with clinical manifestation of acute post streptococcal glomerulonephritis during one year period .
  In addition to meticulous history taking and thorough clinical examination , all the cases will be subjected to the following laboratory investigations :
  Complete blood count on admission, urine analysis, blood urea, serum creatinine, serum albumin, serum cholesterol, urine spot protein creatinine ratio, antistreptolysin O , Erythrocyte sedimentation rate , C-reactive protein and serum complement C3 levels on admission and after 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-27 (Estimated); Primary Completion 2019-06-27 (Estimated); Study Completion 2019-12-27 (Estimated)

PRIMARY OUTCOMES:
number of patients with full recovery or having complication at time of discharge and after 8 week | one year
  serum complementary test by ELISA

REFERENCES:
- [Background] Couser WG. Glomerulonephritis. Lancet. 1999 May 1;353(9163):1509-15. doi: 10.1016/S0140-6736(98)06195-9. PMID 10232333
- [Background] Arimura Y, Muso E, Fujimoto S, Hasegawa M, Kaname S, Usui J, Ihara T, Kobayashi M, Itabashi M, Kitagawa K, Hirahashi J, Kimura K, Matsuo S. Evidence-based clinical practice guidelines for rapidly progressive glomerulonephritis 2014. Clin Exp Nephrol. 2016 Jun;20(3):322-41. doi: 10.1007/s10157-015-1218-8. No abstract available. PMID 27099135
- [Result] Arora P, Kher V, Rai PK, Singhal MK, Gulati S, Gupta A. Prognosis of acute renal failure in children: a multivariate analysis. Pediatr Nephrol. 1997 Apr;11(2):153-5. doi: 10.1007/s004670050247. PMID 9090652
- [Result] Barbiano Di Belgiojoso G, Genderini A, Ferrario F. [Post-infectious glomerulonephritis]. G Ital Nefrol. 2003 Mar-Apr;20(2):184-99. Italian. PMID 12746805
- [Result] Matsukura H, Ohtsuki A, Fuchizawa T, Miyawaki T. Acute poststreptococcal glomerulonephritis mimicking Henoch-Schonlein purpura. Clin Nephrol. 2003 Jan;59(1):64-5. doi: 10.5414/cnp59064. No abstract available. PMID 12572934
- [Result] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Result] Nordstrand A, Norgren M, Holm SE. Pathogenic mechanism of acute post-streptococcal glomerulonephritis. Scand J Infect Dis. 1999;31(6):523-37. doi: 10.1080/00365549950164382. PMID 10680980
- [Result] Kanjanabuch T, Kittikowit W, Eiam-Ong S. An update on acute postinfectious glomerulonephritis worldwide. Nat Rev Nephrol. 2009 May;5(5):259-69. doi: 10.1038/nrneph.2009.44. PMID 19384327